CLINICAL TRIAL: NCT07164859
Title: Safety and Efficacy of Very Short Dual Antiplatelet Therapy Followed by P2Y12 Inhibitor Monotherapy in Older Patients Undergoing Percutaneous Coronary Intervention (SOLOPCI)
Brief Title: Safety and Efficacy of Very Short DAPT in Older Patients Undergoing PCI
Acronym: SOLOPCI
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vincent ROULE (Other)
Responsible Party: Sponsor-Investigator, Vincent ROULE, Principal Investigator, University Hospital, Caen
Organization: University Hospital, Caen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-507545-28-00; 2023-507545-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-25; First posted 2025-09-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease (CAD); Percutaneous Coronary Intervention (PCI); Antiplatelet Therapy; Elderly (People Aged 65 or More)
Keywords: antiplatelet therapy; percutaneous coronary intervention; elderly
MeSH Terms: conditions — Coronary Artery Disease | interventions — 2'-deoxythymidylyl-(3'-5')-2'-deoxyadenosine; Time

STUDY DESIGN:
Intervention Model Description: Multicenter, open label, blinded endpoint assessment, randomized non-inferiority trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard DAPT duration (Active Comparator): Patients assigned to standard DAPT duration will receive DAPT (with aspirin and a P2Y12 inhibitor: ticagrelor, prasugrel or clopidogrel for acute coronary syndrome, or clopidogrel for chronic coronary syndrome) for at least 3 months after randomization or longer and followed by single antiplatelet therapy (aspirin or P2Y12 inhibitor, at the discretion of the local investigator after PCI)
  Interventions: Drug: Standard DAPT duration
- short DAPT (Experimental): Patients assigned to short DAPT will receive DAPT (with aspirin and a P2Y12 inhibitor: ticagrelor, prasugrel or clopidogrel for acute coronary syndrome, or clopidogrel for chronic coronary syndrome) for 7 days (after randomization) followed by P2Y12 inhibitor alone (ticagrelor, prasugrel or clopidogrel as indicated) for 12 months
  Interventions: Drug: short dual antiplatelet therapy (DAPT) duration

INTERVENTIONS:
Drug: short dual antiplatelet therapy (DAPT) duration — patients will receive DAPT for 7 days (after randomization) followed by P2Y12 inhibitor alone
  Arms: short DAPT
Drug: Standard DAPT duration — patients will receive DAPT for at least 3 months after randomization or longer and followed by single antiplatelet therapy
  Arms: standard DAPT duration

SUMMARY:
The goal of this clinical trial is to learn if reducing the duration of dual antiplatelet therapy (DAPT) after percutaneous coronary intervention (short treatment regimen, stopping aspirin at day 7) is as safe and efficient as the standard DAPT duration (standard treatment regimen) in elderly patients ≥ 65 years.

The main questions it aims to answer are:

Does the reduction of the duration of DAPT reduces rates of bleeding without increasing the risk of cardiovascular events? Researchers will compare a short treatment by DAPT (7 days, followed by single antiplatelet therapy) to a standard treatment duration by DAPT (3 to 12 months) after successful percutaneous coronary intervention with ≥ 1 drug-eluting stent.

Participants will:

* Take aspirin for 7 days in one group or 3 to 12 months in another group
* Be contacted by phone at 7 days, 14 days, 21 days, 30 days, 3 months, 6 months and 12 months after hospital discharge
* Keep a diary of any bleeding or cardiovascular events occurring during the study period

DETAILED DESCRIPTION:
While dual antiplatelet therapy (DAPT) is the cornerstone of medical therapy after percutaneous coronary intervention (PCI), its optimal duration is still under debate. DAPT reduces the incidence of thrombotic events but exposes patients to an increased risk of bleeding strongly associated with mortality. Older age is a known predictor of bleeding risk. In the elderly, the duration of DAPT appears to be the most relevant modifiable risk factor.

Bleeding consequences triggered investigations into a further reduction in DAPT duration with the use of the newer generation drug-eluting stent (DES) but none specifically focused on elderly patients. Single antiplatelet therapy (SAPT) using a P2Y12 inhibitor after a short period of DAPT (between 1 and 3 months) has been recently tested in some studies. A meta-analysis focusing on the elderly subgroups (with cut-offs ranging between 65 and 75 years-old) showed similar rates of major bleeding and the composite ischemic endpoint but with a high level of heterogeneity highlighting the need of specific studies in this particular population. A recent large study, including a large proportion of patients ≥ 75 years and comparing SAPT after 1 month of DAPT to DAPT ≥ 3 months, showed a lower incidence of major bleedings while net adverse clinical events and major adverse cardiac events remain non-inferior. In the presence of strong P2Y12 receptor blockade, aspirin provides little additional inhibition of platelet aggregation and inhibition of hemostatic system activation has been reported to be comparable between P2Y12 inhibitor monotherapy and DAPT in healthy subjects. The low thrombogenicity of new coronary devices, potent platelet inhibition with new P2Y12 inhibitors in monotherapy and the potential life-threatening consequences of bleeding which occur mostly in the weeks following PCI support the idea of very short DAPT after PCI in elderly.

The investigators propose a multi-center randomized study to compare the safety and efficacy of very short versus standard-duration DAPT after PCI with DES in elderly patients. The investigators aim to determine whether short DAPT (for 7 days after randomization) followed by SAPT with P2Y12 inhibitor is non inferior to standard-duration DAPT regarding net clinical benefit (a composite of all-cause death, myocardial infarction, stroke, and major bleeding defined by Bleeding Academic Research Consortium (BARC) 3 or 5) at 1 year in elderly patients undergoing PCI for acute or chronic coronary syndrome.

The investigators hypothesized that the very short strategy will be non-inferior to the standard-duration strategy. The very short strategy may allow to further reduce bleedings while maintaining the ischemic risk and may consequently become the default strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 65 years
* Successfully treated with percutaneous coronary intervention (PCI) with ≥ 1 drug-eluting stent (final TIMI 3 flow and visually estimated residual diameter stenosis <30%) for acute coronary syndrome (including ST-elevation myocardial infarction, non-ST-elevation myocardial infarction and unstable angina) or chronic coronary syndrome (elective PCI). Inclusion is possible after the last PCI procedure in staged procedure.
* Randomization must be performed before the discharge from the study site.
* Written informed consent
* Social security affiliated

Exclusion Criteria:

* PCI without drug-eluting stent implantation or with a bioresorbable scaffold
* Planned coronary artery bypass grafting or cardiac surgery
* Any planned surgery within 12 months unless intended antiplatelet therapy could be maintained throughout the peri-surgical period
* Index PCI for stent thrombosis or chronic total occlusion
* Need for oral anticoagulation therapy
* Known hypersensitivity or allergy to aspirin, clopidogrel, ticagrelor or prasugrel
* Use of fibrinolytic therapy within 24 hours of PCI
* Severe renal insufficiency (MDRD creatinine clearance < 30 ml/min/m2) and/or dialysis
* Increased bleeding risk (prior hemorrhagic stroke; stroke < 30 days; brain injury<6 months; history of intracranial tumor or intracranial hemorrhage; internal bleeding<6 weeks; active bleeding; anemia (hemoglobin ≤ 8 g/dl) or thrombocytopenia (platelets < 100 000 G/L); major surgery<3 weeks)
* increased thrombotic risk related to the patient (previous stent thrombosis, ≥ 2 previous myocardial infarction, symptomatic peripheral artery disease, chronic systemic inflammatory disease treated with corticoids or immunosuppressive drug) or the procedure (left main treated, ≥3 stents/treated lesions, total length of stents>60mm, bifurcation lesion with stents in each branch, stenting of the last patent vessel)
* Life expectancy less than 1 year
* Participation in another interventional trial
* Patients considered as vulnerable by the investigators because of medical, psychological or social conditions:

  * Patients with known or discovered severe cognitive impairment
  * Patients with treated or untreated severe psychological or psychiatric conditions
  * Patients with uncorrected severe hearing or visual handicap
  * Patients with addictive alcohol, drug or substance abuse
  * Patients with protective measures (guardianship, tutorship, curatorship)
  * Any other condition considered by the investigators as not warranting informed consent
* patients with poor quality of the downstream territory with diffuse distal coronary disease
* women of childbearing potential: non menopaused -with no menses for 12 months without an alternative medical cause- and not permanently sterilized -hysterectomy, bilateral salpingectomy or bilateral oophorectomy-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
net clinical benefit | 12 months after randomization
  composite of all-cause death, myocardial infarction, stroke and major bleeding BARC 3 or 5

SECONDARY OUTCOMES:
Major or clinically relevant non-major bleeding | 12 months
  Major or clinically relevant non-major bleeding (BARC 2, 3 or 5), non inferiority of the experimental arm tested
Major or clinically relevant non-major bleeding | 12 months
  Major or clinically relevant non-major bleeding (BARC 2, 3 or 5), superiority of the experimental arm tested
Major cardiovascular and cerebrovascular events | 12 months
  a composite of all-cause death, myocardial infarction and stroke, non inferiority of the experimental arm tested
Major bleeding (BARC 3 or 5) | 12 months
  Major bleeding (BARC 3 or 5), superiority of the experimental arm tested

OTHER OUTCOMES:
net clinical benefit | 12 months
  a composite of all-cause death, myocardial infarction, stroke, and major bleeding defined as BARC grade 3 or 5, evaluated as superior or not
all-cause death | 12 months
myocardial infarction | 12 months
  myocardial infarction type 1, 3 or 4b based on the universal definition
Any stroke | 12 months
  Any stroke rates, defined by NeuroARC types 1.a, .b, .c, .d or 1.a.H or 3.a
Intracranial bleeding | 12 months
  Intracranial bleeding rates defined by NeuroARC type 1.a.H, 1.b, 1.c hemorrhagic CNS injury
cardiovascular death | 12 months
  Death of cardiovascular cause (according to ARC-2 definition)
stent thrombosis | 12 months
  stent thrombosis rates (definite or probable, ARC-2 definition)
All-cause hospitalization | 12 months
  hospitalization for any cause, lasting ≥ 24h from the admission to the hospital
Urgent/unplanned symptoms-driven coronary revascularization | 12 months
  Unstable angina leading to coronary revascularization (with percutaneous coronary intervention or coronary artery bypass grafting)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent ROULE, MD, PhD, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No